CLINICAL TRIAL: NCT01061437
Title: A Phase III Randomized Trial of Three Antibiotic Regimens to Eradicate Helicobacter Pylori
Brief Title: S0701, Trial of Three Antibiotic Regimens to Eradicate Helicobacter Pylori (H. Pylori)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0701
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: H. pylori
MeSH Terms: interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Standard 14 day, 3-drug regimen
  Interventions: Drug: PACx14
- Arm 2 (Experimental): Concomitant Therapy - 5 day, 4-drug regimen
  Interventions: Drug: PACMx5
- Arm 3 (Experimental): Sequential Therapy - 10 day, 4-drug regimen
  Interventions: Drug: PAx5/PCMx5

INTERVENTIONS:
Drug: PACx14 — Standard 14 day, 3 drug regimen: lansoprazole, amoxicillin, clarithromycin (PACx14)
  Other Names: Lansoprazole: Prevacid
  Arms: Arm 1
Drug: PACMx5 — Concomitant therapy - 5 day, 4 drug regimen: lansoprazole, amoxicillin, clarithromycin, metronidazole (PACMx5)
  Other Names: Lansoprazole: Prevacid
  Arms: Arm 2
Drug: PAx5/PCMx5 — Sequential Therapy - 10 day, 4-drug regimen: lansoprazole, amoxicillin for 5 days, followed by lansoprazole, clarithromycin and metronidazole for 5 days (PAx5/PCMx5)
  Other Names: Lansoprazole: Prevacid
  Arms: Arm 3

SUMMARY:
The purpose of this study is to compare the effectiveness of three different antibiotic regimens against Helicobacter pylori (H. pylori).

DETAILED DESCRIPTION:
Prevention of gastric cancer through eradication of H. pylori is one of the most promising strategies to reduce the global impact of cancer in the near term. Our long-term goal is to prevent gastric cancer by developing and validating an effective, simple, and low-cost approach to eradication of H. pylori. Our immediate goal, therefore, is to conduct a randomized study to compare the effectiveness of three different drug regimens for H. pylori infection. The three study arms are: Standard therapy - 14 day, 3-drug regimen of Lansoprazole, amoxicillin and clarithromycin (PACx14); Concomitant therapy - 5 day, 4-drug regimen of lansoprazole, amoxicillin, clarithromycin, metronidazole (PACMx5); Sequential therapy - 10 day, 4-drug regimen of lansoprazole, amoxicillin for 5 days, followed by lansoprazole, clarithromycin and metronidazole for 5 days (PAx5/PCMx5).

ELIGIBILITY:
Inclusion Criteria:

* positive Urea Breath Test documenting H. pylori infection
* age 21 - 65 years
* no known allergies to study drugs
* only member of household participating in study
* no known medical conditions (other than H. pylori) that would preclude or require antibiotic therapy
* patients must be willing to discontinue alcohol use for 15 days (maximum duration of treatment plus one day)
* patients must be willing to discontinue use of antacids for duration of study treatment
* patients must not have used proton pump inhibitors (PPI) within 30 days of registration. Patients also must be willing to stop using non-study provided PPIs until the completion of the 6 week follow-up contact.
* patients must not have been treated with antibiotics for H. pylori in the past and must not have taken any other antibiotics within 30 days of registration.
* patients must be willing to return for 2 follow-up visits: 6 weeks after randomization following completion of treatment & 1 year after randomization
* patients must be willing to allow submission of blood for assays of serum markers of bacterial virulence and host genetic susceptibility and environmental factors and provide consent for use of specimens.

Exclusion Criteria:

* current use of anti-retroviral therapy for HIV or AIDS
* diagnosed congestive hear failure
* renal failure requiring dialysis
* diagnosed hepatic failure resulting in hyperbilirubinemia
* any current or prior malignancy except: adequately treated basal or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or Stage II cancer from which the patient has been disease free for 5 years
* pregnancy or nursing mothers

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1859 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To compare 2 experimental antibiotic regimens with a standard 14 day regimen with regard to H. pylori eradication rates at 6 weeks post-randomization. | week 6 post-randomization

SECONDARY OUTCOMES:
Secondary aims will examine infection rates at 1 year, safety and tolerability of these regimens,& potential differential effects among selected groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: E. Robert Greenberg, M.D., Principal Investigator — SWOG Cancer Research Network
Locations (7):
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Universidad del Valle, Cali, Valle del Cauca Department, Colombia
- Fundacion Inciensa, San José, Costa Rica
- Hospital Occidente, Copán, Honduras
- Mexico (2):
  - National Institute for Public Health, Cuernavaca, Morelos
  - Instituto Technologico de Sonora, Obregón, Sonora
- Centro de Investigacion en Demografia y Salud de la Iglesia Merced, León, Nicaragua

REFERENCES:
- [Derived] Morgan DR, Torres J, Sexton R, Herrero R, Salazar-Martinez E, Greenberg ER, Bravo LE, Dominguez RL, Ferreccio C, Lazcano-Ponce EC, Meza-Montenegro MM, Pena EM, Pena R, Correa P, Martinez ME, Chey WD, Valdivieso M, Anderson GL, Goodman GE, Crowley JJ, Baker LH. Risk of recurrent Helicobacter pylori infection 1 year after initial eradication therapy in 7 Latin American communities. JAMA. 2013 Feb 13;309(6):578-86. doi: 10.1001/jama.2013.311. PMID 23403682
- [Derived] Greenberg ER, Anderson GL, Morgan DR, Torres J, Chey WD, Bravo LE, Dominguez RL, Ferreccio C, Herrero R, Lazcano-Ponce EC, Meza-Montenegro MM, Pena R, Pena EM, Salazar-Martinez E, Correa P, Martinez ME, Valdivieso M, Goodman GE, Crowley JJ, Baker LH. 14-day triple, 5-day concomitant, and 10-day sequential therapies for Helicobacter pylori infection in seven Latin American sites: a randomised trial. Lancet. 2011 Aug 6;378(9790):507-14. doi: 10.1016/S0140-6736(11)60825-8. Epub 2011 Jul 21. PMID 21777974
- See also: Click here for more information about the study: S0701, "A Phase III Randomized Trial of Three Antibiotic Regimens to Eradicate Helicobacter Pylori." — http://www.swog.org/